CLINICAL TRIAL: NCT02564302
Title: Effects of Monitored Mindfulness Training on Quality-of-life, Anxiety, and Depression in Patients Awaiting Ablation of Atrial Fibrillation
Brief Title: Effects of Mindfulness on Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newmarket Electrophysiology Research Group Inc (Other)
Responsible Party: Principal Investigator, Pouria Alipour, Research Associate, Newmarket Electrophysiology Research Group Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NERG-03
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
Keywords: PVI; Atrial Fibrillation; MUSE Headband; Mindfulness
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): These patients will not receive a device, but have to fill out a quality of life questionnaire at the time of enrollment and 3 months after their procedure.
- Treatment Group (Experimental): These patients will receive the device. they are expected to use it for at least 5 minutes per day. Patients in this arm will fill out a quality of life questionnaire at the time of enrollment and 3 months after their procedure.
  Interventions: Device: MUSE Headband

INTERVENTIONS:
Device: MUSE Headband — MUSE Headband will help patients with mindfulness.
  Arms: Treatment Group

SUMMARY:
This study aims to investigate the effect of MUSE (R) Headbands on patients with Atrial Fibrillation who is awaiting pulmonary vein isolation ablation procedure. Patients are randomized in 2 arms. The control arm will not be receiving the MUSE headband, whereas the treatment group obtains a device.

Patients from both group will fill out a quality-of-life questionnaire at the time of enrollment and 3 months post PVI. Results from both arms will be evaluated and ultimately the effect of mindfulness using the headband will be evaluated in the aforementioned patient population.

DETAILED DESCRIPTION:
Background:

Atrial fibrillation is the most common arrhythmic disorder and ablation of AF has become an important part of AF treatment. AF is associated with a large number of somatic symptoms like chest pain, fatigue, lightheadedness, palpitations, physical limitations, shortness of breath, irregular rhythm and heart rate but also with psychological comorbidities such as anxiety and depression [1]. In recent years, the severity of these comorbidities has become more apparent in AF patients. For instance, Sears and colleagues found a positive correlation between the number of AF symptoms reported and the number of negative emotions experienced [2]. Since there is prospective data on the effects of AF ablation on long term mortality and morbidity, reduction of AF related symptoms and improvement of quality of life (QoL) is still a major goal of AF ablation [3,4].

Mindful meditation (MM) is a basic form of meditation that involves focusing on one thing internally or externally. Being fully present in the moment is the goal of MM. Practicing MM teaches relaxation and concentration on experiencing bodily sensations such as breathing patterns. Mindfulness is independent of environmental stimuli; it is a state of mind that can be achieved at any time [5]. Studies show that, with practice, this form of meditation can provide both long- and short-term positive effects with respect to reduction in anxiety and depression[6,7]. Immediate and transferable benefits for AF patients include self-regulated attention, heightened perception of internal states, reduced stress and anxiety symptoms, and increased overall well-being.

Mindfulness training can heighten meta-cognitive processing, which can improve a person's ability to control adverse thoughts and feelings. Consistent mindful meditation training can induce neuroplasticity[7,8].

The amygdala is a crucial brain structure that is hyperactive during perceived stressful conditions [8]. Being able to utilize skills to control emotions in stressful situations will be beneficial in controlling psychological hyperactivity. Studies show after mindful-attention training there is a decrease in amygdala activity even when in a non-meditative state [6]. This is proof that skills obtained during meditation have lasting positive neural effects. In another study, Holzel et al. found that after eight weeks of MM training, there was a significant correlation between a decrease in subjective stress and a decrease in amygdala's gray matter density. Therefore, a reduction in stress output is positively correlated with gray matter density. MM training induces brain changes in the amygdala and resting state connectivity, which have impacts on cognition such as an increase in attentional control and executive function [9].

Neurofeedback training (NFT) is a method where participants are hooked up to an EEG which allows participants to see how active their brain is and monitor neural changes in real-time. NFT is proven to significantly enhance the positive effects of MM training and have a positive effect on depression[10,11].

The present study is going to investigate the psychological and physiological benefits of mindful meditation (MM) training in patients with atrial fibrillation (AF) using a system for real-time-neurofeedback.

Rationale for study design:

Although there is growing evidence that there might also positive prognostic effects especially on stroke risk [12,13] treatment of AF related symptoms is still one of the major targets of AF ablation. Lakkireddy and colleagues showed that yoga could improve symptoms and QoL as well as anxiety and depression scores [14] in AF patients, illustrating that alternative therapy can be highly effective in AF and be a valuable addition to somatic therapy like AF-ablation.

In this study investigators want to investigate the effects of mindfulness meditation that is supported by the MUSE™ headband which is a device that provides neurofeedback during the meditation. This way investigators seek not only to improve the effects of the meditation but also will be able to monitor therapy compliance via the implemented software.

Since patients with AF are a very heterogeneous group and AF burden, comorbidities as well as symptom perception can differ significantly investigators chose to investigate the less diverse group of patients with symptomatic AF that are scheduled for AF ablation. By applying prospective randomization investigators avoid the risk of a significant bias in baseline patient characteristics and comorbidities.

Study design and aims:

A total number of 60 patients waiting for an AF ablation for symptomatic AF will be included into this prospective, randomized pilot study. All patients will undergo assessment of QoL, anxiety and depression using 3 self-reporting scales for QoL, anxiety and depression at baseline and after 12 weeks. The scales are listed in Appendix A.

At baseline patients will be 1:1 randomized to be either part of the intervention (Group 1) or control (Group 2) group. Patients in Group 1 will be supplied with the MUSE™ headband (InteraXon Inc., Toronto, Canada) that is a tool for mindfulness meditation with neurofeedback. Patients in Group 2 will not undergo any study-related treatment.

The aim of this study will be to investigate the effects of mindfulness meditation with neurofeedback on QoL, anxiety and depression in patients awaiting AF ablation. The results of the study will also be the basis of future studies further investigating the

Statistical analysis:

The primary endpoint will be expressed as mean or median test result where applicable. The secondary endpoint will be measured by the individual duration of use of the device in group 1. The Shapiro-Wilks-test will be used to test for normality of distribution and the Mann-Whitney-U test will be applied for comparison of means.

Study-timeline and Budget:

Our institution is a high volume centre for AF ablations that performs 300-350 procedures per year. Because of the non-invasive character of the MUSE-device investigators expect a high recruitment rate and plan to complete enrollment of the 60 patients within 6 months. With a follow-time of 3 months investigators expect to complete patient inclusion and follow-up after 9 months. Data analysis will take approximately 4 weeks resulting in a total study duration of 10 months.

InteraXon Inc. will provide 30 MUSE™ headbands for the study time.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* symptomatic persistent or paroxysmal AF awaiting ablation of AF

Exclusion Criteria:

* Known Anxiety and Depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 12 weeks
  patients in both arms will fill out a questionnaire for QoL 12 weeks after their ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Study Director — Newmarket Electrophysiology Research Group
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada